CLINICAL TRIAL: NCT06905483
Title: Comparative Effects of Triple Inhaled Therapy With Budesonide/Glycopyrronium/Formoterol Versus Fluticasone Furoate/Umeclidinium/Vilanterol on Small Airway Disease in COPD Patients: A Randomized Crossover Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Narongkorn Saiphoklang, MD, Associate Professor, Thammasat University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MTU-EC-IM-5-271/67
Record Dates: First submitted 2025-03-22; First posted 2025-04-01 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease (COPD); Small Airway Disease; Triple Therapy; Lung Function
Keywords: COPD; chronic obstructive pulmonary disease; small airway disease; triple inhaled therapy; Budesonide/Glycopyrronium/Formoterol; Fluticasone Furoate/Umeclidinium/Vilanterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; fluticasone furoate

STUDY DESIGN:
Intervention Model Description: This study is a randomized crossover study. COPD patients aged 40 years or older with stable disease are included. Each patient receives four weeks of treatment with either BGF or FUV followed by a one-week washout period, and then four weeks of treatment with the other drug. Respiratory symptoms, pulmonary function, and safety are assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Budesonide/Glycopyrronium/Formoterol (BGF) (Experimental): BGF (160/7.2/5 mcg) 2 inhalations, twice daily for 4 weeks
  Interventions: Drug: Budesonide/Glycopyrronium/Formoterol (BGF); Drug: Fluticasone Furoate/Umeclidinium/Vilanterol (FUV)
- Fluticasone Furoate/Umeclidinium/Vilanterol (FUV) (Active Comparator): FUV (100/62.5/25 mcg) 1 inhalation, once daily for 4 weeks
  Interventions: Drug: Budesonide/Glycopyrronium/Formoterol (BGF); Drug: Fluticasone Furoate/Umeclidinium/Vilanterol (FUV)

INTERVENTIONS:
Drug: Budesonide/Glycopyrronium/Formoterol (BGF) — Each patient received 4 weeks of treatment with either BGF or FUV followed by a 1-week washout period, and then 4 weeks of treatment with the other drug.
  Other Names: Breztri
Drug: Fluticasone Furoate/Umeclidinium/Vilanterol (FUV) — Each patient received 4 weeks of treatment with either BGF or FUV followed by a 1-week washout period, and then 4 weeks of treatment with the other drug.
  Other Names: Trelegy

SUMMARY:
The goal of this clinical trial is to determine if triple inhaled therapy with Budesonide/Glycopyrronium/Formoterol (BGF) and Fluticasone Furoate/Umeclidinium/Vilanterol (FUV) are effective in treating patients with stable chronic obstructive pulmonary disease (COPD). It will also assess the safety of both drugs.

The main questions it aims to answer are:

* Does BGF demonstrate a comparable effect to FUV in COPD participants?
* What medical problems do participants experience when taking BGFand FUV?

DETAILED DESCRIPTION:
This study is a randomized crossover study. COPD patients aged 40 years or older with stable disease are included. Each patient receives four weeks of treatment with either BGF or FUV followed by a one-week washout period, and then four weeks of treatment with the other drug. Respiratory symptoms are assessed using modified Medical Research Council (mMRC) dyspnea scale and COPD Assessment Test (CAT). Pulmonary function is assessed by spirometry with bronchodilator testing, and adverse events were recorded. Spirometry data, including forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and forced expiratory flow at 25-75% of FVC (FEF25-75) are also collected. Impulse oscillometry (IOS) is also performed, with results reported as R5, R20, R5-R20, X5, Fres, and Ax.

ELIGIBILITY:
Inclusion Criteria:

* COPD diagnosis confirmed by spirometry (post-bronchodilator FEV1/FVC < 70%)
* Aged 40-80 years
* Smoking 10 pack-years or more
* Postbronchodilator FEV1 < 80%

Exclusion Criteria:

* History of COPD exacerbation within 3 months
* Asthma, bronchiectasis, pulmonary fibrosis
* Inability to perform spirometry, impulse oscillometry, or 6-minute walk test
* Pregnant or breastfeeding women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-01-28 (Actual)

PRIMARY OUTCOMES:
Changes in airway resistance at 5 Hz (R5) on COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in R5 assessed by impulse oscillometry (IOS), reported as kPa/L/s and percent predicted value.
Changes in airway resistance at 20 Hz (R20) on COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in R20 assessed by impulse oscillometry (IOS), reported as kPa/L/s and percent predicted value.
Difference of airway resistance between 5 Hz and 20 Hz (R5-R20) on COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in R5-R20 assessed by impulse oscillometry (IOS), reported as kPa/L/s.
Reactance at 5 Hz (X5) on COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in X5 assessed by impulse oscillometry (IOS), reported as kPa/L/s.

SECONDARY OUTCOMES:
Changes in forced expiratory volume in 1 second (FEV1) in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in FEV1 assessed by spirometry, reported as liter (L) and percent predicted value.
Changes in forced vital capacity (FVC) in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in FVC assessed by spirometry, reported as liter (L) and percent predicted value.
Changes in FEV1/FVC ratio in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in FEV1/FVC ratio assessed by spirometry, reported as percent.
Changes in forced expiratory flow at 25-75% of FVC (FEF25-75) in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in FEF25-75 assessed by spirometry, reported as liter/second (L/s) and percent predicted value.
Changes in modified Medical Research Council dyspnea scale in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in this dyspnea scale are reported in points, with a minimum range of 0 and a maximum of 5. Higher scores indicate more symptoms.
Changes in COPD assessment test score in COPD patients | From enrollment to the end of treatment at 8 weeks
  Changes in this score are reported in points, with a minimum range of 0 and a maximum of 40. Higher scores indicate more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Narongkorn Saiphoklang, MD, Principal Investigator — Thammasat University Faculty of Medicine
Locations (1):
- Narongkorn Saiphoklang, Pathum Thani, Changwat Pathum Thani, Thailand

IPD SHARING:
Plan to Share IPD: Yes
IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and documents will be available for sharing immediately after publication for a period of 2 years.
Access Criteria: All researchers will be able to access the IPD and supporting information via the repository website without restriction.

REFERENCES:
- [Result] Usmani O, Li G, De Backer J, Sadafi H, Wu L, Marshall J. Modeled small airways lung deposition of two fixed-dose triple therapy combinations assessed with in silico functional respiratory imaging. Respir Res. 2023 Sep 23;24(1):226. doi: 10.1186/s12931-023-02534-y. PMID 37742015
- [Result] Usmani OS, Scichilone N, Mignot B, Belmans D, Van Holsbeke C, De Backer J, De Maria R, Cuoghi E, Topole E, Georges G. Airway Deposition of Extrafine Inhaled Triple Therapy in Patients with COPD: A Model Approach Based on Functional Respiratory Imaging Computer Simulations. Int J Chron Obstruct Pulmon Dis. 2020 Oct 7;15:2433-2440. doi: 10.2147/COPD.S269001. eCollection 2020. PMID 33116458
- [Result] Bremner PR, Birk R, Brealey N, Ismaila AS, Zhu CQ, Lipson DA. Single-inhaler fluticasone furoate/umeclidinium/vilanterol versus fluticasone furoate/vilanterol plus umeclidinium using two inhalers for chronic obstructive pulmonary disease: a randomized non-inferiority study. Respir Res. 2018 Jan 25;19(1):19. doi: 10.1186/s12931-018-0724-0. PMID 29370819
- [Result] Bansal S, Anderson M, Anzueto A, Brown N, Compton C, Corbridge TC, Erb D, Harvey C, Kaisermann MC, Kaye M, Lipson DA, Martin N, Zhu CQ, Papi A. Single-inhaler fluticasone furoate/umeclidinium/vilanterol (FF/UMEC/VI) triple therapy versus tiotropium monotherapy in patients with COPD. NPJ Prim Care Respir Med. 2021 May 25;31(1):29. doi: 10.1038/s41533-021-00241-z. PMID 34035312
- [Result] Lipson DA, Barnacle H, Birk R, Brealey N, Locantore N, Lomas DA, Ludwig-Sengpiel A, Mohindra R, Tabberer M, Zhu CQ, Pascoe SJ. FULFIL Trial: Once-Daily Triple Therapy for Patients with Chronic Obstructive Pulmonary Disease. Am J Respir Crit Care Med. 2017 Aug 15;196(4):438-446. doi: 10.1164/rccm.201703-0449OC. PMID 28375647
- [Result] Maneechotesuwan K, Sawatdee S, Srichana T. In Vitro Analysis of Aerodynamic Properties and Co-Deposition of a Fixed-Dose Combination of Fluticasone Furoate, Umeclidinium Bromide, and Vilanterol Trifenatate. Pharmaceutics. 2024 Oct 18;16(10):1334. doi: 10.3390/pharmaceutics16101334. PMID 39458663
- [Result] Martinez FJ, Rabe KF, Ferguson GT, Wedzicha JA, Trivedi R, Jenkins M, Darken P, Aurivillius M, Dorinsky P. Benefits of budesonide/glycopyrrolate/formoterol fumarate (BGF) on symptoms and quality of life in patients with COPD in the ETHOS trial. Respir Med. 2021 Aug-Sep;185:106509. doi: 10.1016/j.rmed.2021.106509. Epub 2021 Jun 18. PMID 34171789
- [Result] Ishiura Y, Fujimura M, Ohkura N, Hara J, Kasahara K, Ishii N, Sawai Y, Shimizu T, Tamaki T, Nomura S. Triple Therapy with Budesonide/Glycopyrrolate/Formoterol Fumarate Improves Inspiratory Capacity in Patients with Asthma-Chronic Obstructive Pulmonary Disease Overlap. Int J Chron Obstruct Pulmon Dis. 2020 Feb 5;15:269-277. doi: 10.2147/COPD.S231004. eCollection 2020. PMID 32103926
- [Result] Rabe KF, Martinez FJ, Singh D, Trivedi R, Jenkins M, Darken P, Aurivillius M, Dorinsky P. Improvements in lung function with budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler versus dual therapies in patients with COPD: a sub-study of the ETHOS trial. Ther Adv Respir Dis. 2021 Jan-Dec;15:17534666211034329. doi: 10.1177/17534666211034329. PMID 34428980
- [Result] Ferguson GT, Rabe KF, Martinez FJ, Fabbri LM, Wang C, Ichinose M, Bourne E, Ballal S, Darken P, DeAngelis K, Aurivillius M, Dorinsky P, Reisner C. Triple therapy with budesonide/glycopyrrolate/formoterol fumarate with co-suspension delivery technology versus dual therapies in chronic obstructive pulmonary disease (KRONOS): a double-blind, parallel-group, multicentre, phase 3 randomised controlled trial. Lancet Respir Med. 2018 Oct;6(10):747-758. doi: 10.1016/S2213-2600(18)30327-8. Epub 2018 Sep 16. PMID 30232048
- [Result] Usmani O, Roche N, Wahab E, Israel S, Jenkins M, Trivedi R, Dorinsky P, Aurivillius M. A scintigraphy study of budesonide/glycopyrrolate/formoterol fumarate metered dose inhaler in patients with moderate-to-very severe chronic obstructive pulmonary disease. Respir Res. 2021 Oct 7;22(1):261. doi: 10.1186/s12931-021-01813-w. PMID 34620167
- [Result] Bickel S, Popler J, Lesnick B, Eid N. Impulse oscillometry: interpretation and practical applications. Chest. 2014 Sep;146(3):841-847. doi: 10.1378/chest.13-1875. PMID 25180727
- [Result] McNulty W, Usmani OS. Techniques of assessing small airways dysfunction. Eur Clin Respir J. 2014 Oct 17;1. doi: 10.3402/ecrj.v1.25898. eCollection 2014. PMID 26557240
- [Result] Lazarinis N, Fouka E, Linden A, Bossios A. Small airways disease in chronic obstructive pulmonary disease. Expert Rev Respir Med. 2024 Jul;18(7):539-552. doi: 10.1080/17476348.2024.2380070. Epub 2024 Jul 24. PMID 39046133
- [Result] Singh D, Long G, Cancado JED, Higham A. Small airway disease in chronic obstructive pulmonary disease: insights and implications for the clinician. Curr Opin Pulm Med. 2020 Mar;26(2):162-168. doi: 10.1097/MCP.0000000000000637. PMID 31688242
- [Result] Verleden SE, Hendriks JMH, Snoeckx A, Mai C, Mentens Y, Callebaut W, De Belie B, Van Schil PE, Verplancke V, Janssens A, Jacob J, Pakzad A, Conlon TM, Guvenc G, Yildirim AO, Pauwels P, Koljenovic S, Kwakkel-Van Erp JM, Lapperre TS. Small Airway Disease in Pre-Chronic Obstructive Pulmonary Disease with Emphysema: A Cross-Sectional Study. Am J Respir Crit Care Med. 2024 Mar 15;209(6):683-692. doi: 10.1164/rccm.202301-0132OC. PMID 38055196
- [Result] Sudi A, Santa B, Horvath A, Tomisa G, Abonyi-Toth Z, Rokszin G, Eszes N, Muller V, Tamasi L. The Real-World Efficacy of Fixed Triple Inhalation Therapy in the Treatment of Moderate COPD Patients (RATIONALE Study). Int J Chron Obstruct Pulmon Dis. 2024 Aug 28;19:1943-1955. doi: 10.2147/COPD.S474354. eCollection 2024. PMID 39219564